CLINICAL TRIAL: NCT06008379
Title: A Phase 1/2 Dose Escalation and Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of 7MW3711 in Subjects With Advanced Solid Tumors
Brief Title: A Study of 7MW3711 in Subjects With Advanced Solid Tumors
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 7MW3711-2023-CP102
Record Dates: First submitted 2023-08-07; First posted 2023-08-23 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Advanced Solid Tumor
MeSH Terms: interventions — Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dose escalation and dose expansion (Experimental): all subjects enrolled in the part of dose escalation and dose expansion will receive 7MW3711 by introvenous infusion
  Interventions: Drug: 7MW3711 for injection
- cohort expansion (Experimental): all subjects enrolled in the part of cohort expansion will be treated by 7MW3711 will receive 7MW3711 by introvenous infusion
  Interventions: Drug: 7MW3711 for injection

INTERVENTIONS:
Drug: 7MW3711 for injection — IV administration of 7MW3711, Q3W, 3 weeks a cycle
  Arms: dose escalation and dose expansion
Drug: 7MW3711 for injection — IV administration of 7MW3711, the dosage regimen including dosage and dosing frequency for cohort expansion is conformed on basis of the data in part 1
  Arms: cohort expansion

SUMMARY:
7MW3711 is a antibody-drug conjugate(ADC) drected to a target wildly expressed on solid tumors. This is an open-label, multicenter, phase 1/2 study to evaluate the Safety, Tolerability, Pharmacokinetics, and Efficacy of 7MW3711 in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
Two parts are included in this study. The part of dose escalation and dose expansion(part 1) will enrolled subjects with advanced solid tumors and is to evaluate the safety and tolerability and to determine the maximum tolerated dose and/or the recommend pahse 2 dose(RP2D) of 7MW3711 in subjects with advanced solid tumors.

The part of cohort expansion(part 2) will enrolled subejcts with selected advanced solid tumors and is to assess the preliminary efficacy of 7MW3711 in selected advanced solid tumors.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
* Life expectancy of at least 3 months as assessed by the Investigator.
* Part 1: Histologically or cytologically confirmed locally advanced or metastatic solid tumor, progressive after last treatment received and who progressed on or after standard therapies or intolerant to approved therapies or who lack of effient standard therapies; part 2: Histologically or cytologically confirmed locally advanced or metastatic selected advanced solid tumors having progressed after at least one line of standard systermic therapy or intolerate standard therapies.
* An archival tumor tissue sample(formalin-fixed paraffin-embedded (FFPE) tumor tissue block or at least 5 unstained slides) or a fresh tissue sample should be provided. If the tissue sample cannot be provided during dose escalation, enrollment into the study is allowed after discussion with the Investigator
* Measurable or evaluable disease by RECIST v1.1.
* Have adequate hematopoietic, renal and hepatic functions.
* Men or women willing to use adequate contraceptive measures throughout the study

Exclusion Criteria:

* Have other prior malignancies within 3 years before the first administration.
* Known central nervous system metastatic disease or carcinomatous meningitis except for treated and stable brain metastases.
* Have significant, uncontrolled, or active cardiovascular disease.
* Known history of COPD, or intestinal lung disease, or other respiratory diseases requring inpatient treatments within 4 weeks prior to first administration.
* Have adverse events due to prior antitumor therapy not resolved to grade 1 or lower by NCI CTCAE V5.0.
* have active infections requiring treatment within 14 weeks; have infection of HIV, active infection of HCV and HBV.
* Prior treatment with an antibody drug conjugate (ADC) that consists of an topoisomerase I inhibitor.
* Prior treatment with B7-H3 targeted agents.
* have received chemotherapy, immunotherapy, curative radiation within 3 weeks prior to the first administration or targeted molecular within 2 weeks prior to first administration. have received Chinese patent medicine or Chinese herbs of anti-tumor indications within 1 weeks prior to the first administration.
* Have received any systemic immunosuppressants within 2 weeks prior to the first administration except for topical corticosteroids.
* Have received any other investigational drugs or medical device within 4 weeks prior to the first administration.
* History of drug abuse including narcotic and psychiatric drugs within 12 months prior to screening.
* Pregnant, or nursing females

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 164 (Estimated)
Dates: Start 2023-08-28 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2026-01-30 (Estimated)

PRIMARY OUTCOMES:
evaluation of the incidence of adverse events (AEs) (part 1) | approximately up to 16 cycles, 21 days a cycle
  Incidence and seriousness of adverse events (AEs) and serious adverse events (SAEs) by CTCAE version 5.0.
Identification of the MTD and /or RP2D of 7MW3711(part 1) | from Day1 to Day21 in cycle1 of part 1
Overall response rate (ORR) evaluated by investigators based on RECIST version 1.1 in selected solid tumors. (part 2) | approximately up to 2 years
  ORR:defined as the proportion of patients who achieved a best overall response of completeresponse (CR) or partial response (PR)

SECONDARY OUTCOMES:
evaluation of PK parameters of 7MW3711 | approximately up to 2 years
  Maximum observed concentration(Cmax)
evaluation of PK parameters of 7MW3711 | approximately up to 2 years
  the time to Cmax(tmax)
evaluation of PK parameters of 7MW3711 | approximately up to 2 years
  half-live(t1/2)
evaluation of PK parameters of 7MW3711 | approximately up to 2 years
  Area under the concentration-time curve(AUC)
overall response rate (ORR) (part1) | approximately up to 1 years
  ORR:defined as the proportion of patients who achieved a best overall response of completeresponse (CR) or partial response (PR) based on RECIST version 1.1.
disease control rate(DCR) | approximately up to 2 years
  DCR:defined as the proportion of subjects with CR, PR, and SD based on RECIST 1.1 criteria
progression-free survival(PFS) | approximately up to 2 years
  PFS:defined as time from the date of first administration to the date of first documented disease progression based on RECIST 1.1 criteria, or death due to any cause, whichever occurs first
time to response (TTR) | approximately up to 2 years
  TTR:defined as time from the date of first administration to the date of first documented CR or PR
evaluation of the immunogenicity of 7MW3711 | approximately up to 2 years
  Frequency and percentage of subjects with positive anti-drug antibody after being treated by 7MW3711.
evaluation of the incidence of adverse events (AEs) (part 2) | approximately up to 2 years
  Incidence and seriousness of adverse events (AEs) and serious adverse events (SAEs) by CTCAE version 5.0.

CONTACTS AND LOCATIONS:
Locations (5):
- China (5):
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - The Lung Cancer Center of Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No